CLINICAL TRIAL: NCT01490125
Title: A Multicenter, Randomized, Blinded, Double-dummy, Placebo-controlled, 3-period Cross-over Study to Evaluate the Effect of QVA149 on Patient Reported Dyspnea in Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD), Using Tiotropium as an Active Control
Brief Title: The Effect of QVA149 on Patient Reported Dyspnea in Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Acronym: BLAZE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149A2322; 2011-000229-63 (EudraCT Number)
Record Dates: First submitted 2011-11-15; First posted 2011-12-12 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Dyspnea; QVA149; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — indacaterol-glycopyrronium combination; Tiotropium Bromide; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- QVA149 + placebo to tiotropium (Experimental): Participants received QVA149 plus placebo to tiotropium during 1 of 3 treatment periods, once a day for 6 weeks. Participants were provided with a salbutamol/albuterol inhaler to use as rescue medication.
  Interventions: Drug: QVA149; Drug: Placebo to tiotropium; Drug: Salbutamol/albuterol
- Tiotropium + placebo to QVA149 (Active Comparator): Participants received tiotropium 18 μg plus placebo to QVA149 during 1 of 3 treatment periods once a day for 6 weeks. Participants were provided with a salbutamol/albuterol inhaler to use as rescue medication.
  Interventions: Drug: Tiotropium; Drug: Placebo to QVA149; Drug: Salbutamol/albuterol
- Placebo (Placebo Comparator): Participants received placebo to QVA149 plus placebo to tiotropium during 1 of 3 treatment periods once a day for 6 weeks. Participants were provided with a salbutamol/albuterol inhaler to use as rescue medication.
  Interventions: Drug: Placebo to QVA149; Drug: Placebo to tiotropium; Drug: Salbutamol/albuterol

INTERVENTIONS:
Drug: QVA149 — QVA149 110/50 μg hard non-gelatin capsule, inhalation/blister once a day via SDDPI
  Arms: QVA149 + placebo to tiotropium
Drug: Tiotropium — Tiotropium 18 ug hard gelatin capsule, inhalation/ blister once a day via HandiHaler® device
  Arms: Tiotropium + placebo to QVA149
Drug: Placebo to QVA149 — Placebo 0 mg hard non-gelatin capsule, inhalation/ blister once a day via SDDPI
  Arms: Placebo; Tiotropium + placebo to QVA149
Drug: Placebo to tiotropium — Placebo 0 mg hard gelatin capsule, inhalation/ blister once a day via HandiHaler® device
  Arms: Placebo; QVA149 + placebo to tiotropium
Drug: Salbutamol/albuterol — salbutamol/albuterol (containing CFC-free propellant -HFA 134a) inhaler used as rescue medication when needed.

SUMMARY:
This study assessed the effect of QVA149 on patient-reported dyspnea in moderate to severe Chronic Obstructive Pulmonary Disease (COPD) patients.

DETAILED DESCRIPTION:
This study used a multi-center, randomized, blinded, double-dummy placebo controlled, three-period crossover design to assess the effect of once daily QVA149 q.d vs. placebo and tiotropium 18 μg q.d. in terms of patient reported dyspnea as assessed by Baseline Dyspnea Index (BDI)/Transient Dyspnea Index (TDI)(SAC version) in patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe stable chronic obstructive pulmonary disease
* Smoking history of 10 pack years
* Post-bronchodilator Forced Expiratory Volume in 1 second (FEV1) between 30 - 80%
* Patients must be able to use computer mouse and display
* mMRC grade>2

Exclusion Criteria:

* Patients with a history of long QT syndrome
* Patients with Type I or uncontrolled Type II diabetes
* Patients who have had a COPD exacerbation or respiratory tract infection within 6 weeks prior to screening
* Patients with any history of asthma
* Patients with pulmonary lobectomy, lung volume reduction surgery, or lung transplantation
* Patients with concomitant pulmonary disease
* Patients requiring long term oxygen therapy (>15 h a day)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- Belgium (8):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Gilly
  - Novartis Investigative Site, Jambes
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Ostend
  - Novartis Investigative Site, Wavre
- Canada (6):
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Laval, Quebec
  - Novartis Investigative Site, Mirabel, Quebec
  - Novartis Investigative Site, Saint-Charles-Borromée, Quebec
- Germany (14):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Potsdam, Germany
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rheine
  - Novartis Investigative Site, Rüdersdorf
- Spain (5):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Mérida, Badajoz
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Ponferrada, Leon
  - Novartis Investigative Site, Madrid, Madrid
- United Kingdom (5):
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Portsmouth

REFERENCES:
- [Derived] Mahler DA, Decramer M, D'Urzo A, Worth H, White T, Alagappan VK, Chen H, Gallagher N, Kulich K, Banerji D. Dual bronchodilation with QVA149 reduces patient-reported dyspnoea in COPD: the BLAZE study. Eur Respir J. 2014 Jun;43(6):1599-609. doi: 10.1183/09031936.00124013. Epub 2013 Oct 31. PMID 24176997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 247 patients were randomized. Of these 247, one patient was misrandomized, did not receive study treatment and was excluded from any analysis set. Of 246 patients, 191 completed the study. This is a crossover study; therefore, participants are counted more than once depending on their dosing sequences.
Pre-assignment Details: Participants were randomized to 1 of 6 treatment sequences to receive 1 of 3 treatment combinations; then, crossed to the other 2 possible treatment combinations for a total of 3 treatment periods. Each treatment combination period was followed by a 14 day washout.
Groups:
- QVA149+ Placebo+ Tiotropium: Participants were randomized to sequence QVA149 + placebo + tiotropium.
- QVA149+ Tiotropium+ Placebo: Participants were randomized to sequence QVA149 + tiotropium + placebo.
- Placebo + QVA149 + Tiotropium: Participants were randomized to sequence placebo + QVA149 + tiotropium
- Placebo+ Tiotropium + QVA149: Participants were randomized to sequence placebo + tiotropium + QVA149
- Tiotropium + QVA149+ Placebo: Participants were randomized to sequence tiotropium + QVA149 + placebo
- Tiotropium + Placebo +QVA149: Participants were randomized to sequence tiotropium + placebo + QVA149
Period: Period I
Arm/Group | QVA149+ Placebo+ Tiotropium | QVA149+ Tiotropium+ Placebo | Placebo + QVA149 + Tiotropium | Placebo+ Tiotropium + QVA149 | Tiotropium + QVA149+ Placebo | Tiotropium + Placebo +QVA149
Started | 43 | 42 | 41 | 38 | 40 | 42
Completed | 37 | 37 | 37 | 33 | 36 | 37
Not Completed | 6 | 5 | 4 | 5 | 4 | 5
Not completed — Adverse Event | 4 | 1 | 1 | 3 | 2 | 4
Not completed — Protocol Violation | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 1 | 2 | 1
Period: Period II
Arm/Group | QVA149+ Placebo+ Tiotropium | QVA149+ Tiotropium+ Placebo | Placebo + QVA149 + Tiotropium | Placebo+ Tiotropium + QVA149 | Tiotropium + QVA149+ Placebo | Tiotropium + Placebo +QVA149
Started | 37 | 37 | 37 | 33 | 36 | 37
Completed | 34 | 33 | 34 | 30 | 32 | 35
Not Completed | 3 | 4 | 3 | 3 | 4 | 2
Not completed — Adverse Event | 2 | 3 | 2 | 2 | 4 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Period III
Arm/Group | QVA149+ Placebo+ Tiotropium | QVA149+ Tiotropium+ Placebo | Placebo + QVA149 + Tiotropium | Placebo+ Tiotropium + QVA149 | Tiotropium + QVA149+ Placebo | Tiotropium + Placebo +QVA149
Started | 34 | 33 | 34 | 30 | 32 | 35
Completed | 31 | 32 | 34 | 28 | 31 | 35
Not Completed | 3 | 1 | 0 | 2 | 1 | 0
Not completed — Adverse Event | 3 | 1 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: One misrandomized participant did not receive study treatment, was discontinued and not included in the full analysis set used for demographics.
Groups:
- All Participants: All participants who entered the study and were randomized to any of the 3 treatment combinations: QVA149 plus placebo to tiotropium; tiotropium plus placebo to QVA149 or placebo to QVA149 plus placebo to tiotropium.
Arm/Group | All Participants
Number analyzed (Participants) | 246
Age Continuous [Mean (Standard Deviation); unit: years] | 62.8 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 173

OUTCOME MEASURES:

1. Primary Outcome: Total Total Transient Dyspnea Index (TDI) Score After 6 Weeks of Treatment QVA149 Compared to Placebo
Description: Total Transient Dyspnea Index (TDI) is part of the BDI/TDI questionnaire where participants indicated whether they improved or deteriorated since their Baseline Dyspnea Index (BDI). The BDI and TDI each had 3 domains: activities, tasks, and effort. BDI domains were rated from 0 (very severe) to 4 (none) and the rates summed for the total BDI score ranging from 0 to 12; the lower the score the worse the severity of dyspnea. TDI domains were rated from -6 (major deterioration) to 6 (major improvement) and the rates summed for the total TDI score ranging from -18 to 18. However, to ensure comparability with the TDI paper version, all TDI values were divided by 2 before the analysis. If data was missing or insufficient for any one of the domains a BDI/TDI was calculated. BDI = Baseline Dyspnea Index taken 75 min prior to the first dose in each treatment period. TDI = Transition Dyspnea Index taken after 6 weeks of treatment 75 min prior to the last dose in each treatment period.
Time Frame: Baseline and 6 weeks
Population: The analysis set includes all randomized patients who received at least one dose of study drug and for whom data are available. Data was analyzed according to the treatment they were randomized. In this cross-over design the number of patients on each treatment does not add up to the total number of patients.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | QVA149 + Placebo to Tiotropium | Tiotropium + Placebo to QVA149 | Placebo
Number analyzed (Participants) | 220 | 0 | 218
Units on a scale
  BDI | 7.34 (2.033) |  | 7.33 (2.206)
  TDI | 0.98 (2.666) |  | -0.38 (2.308)

2. Secondary Outcome: Total Total Transient Dyspnea Index (TDI) Score After 6 Weeks of Treatment QVA149 Compared to Tiotropium
Description: as for outcome 1
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | QVA149 + Placebo to Tiotropium | Tiotropium + Placebo to QVA149 | Placebo
Number analyzed (Participants) | 220 | 217 | 0
Units on a scale
  BDI | 7.34 (2.033) | 7.31 (2.199) |
  TDI | 0.98 (2.666) | 0.47 (2.184) |

3. Secondary Outcome: Standardized Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) 5min-4h After First Dose and 6 Weeks of Treatment With QVA149 Compared to Placebo and Tiotropium
Description: Forced Expiratory Volume in 1 second (FEV1) was measured with spirometry conducted according to internationally accepted standards. Measurements were taken at 5 min- 4hr post-dose of day 1 and week 6. The standardized FEV1 Area under the curve (AUC) was calculated as the sum of trapezoids divided by the length of time.
Time Frame: 5min-4hr at day 1 and week 6 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 + Placebo to Tiotropium | Tiotropium + Placebo to QVA149 | Placebo
Number analyzed (Participants) | 223 | 220 | 218
Liters
  Day 1 (n=220,219,2117) | 1.564 (0.0082) | 1.496 (0.0082) | 1.352 (0.0082)
  Week 6 (n=205,209,206) | 1.636 (0.0122) | 1.529 (0.0122) | 1.302 (0.0122)

4. Secondary Outcome: Standardized Forced Vital Capacity (FVC) Area Under the Curve (AUC) 5min-4 Hrs After First Dose and 6 Weeks of Treatment With QVA149 Compared to Placebo and Tiotropium
Description: Forced Vital Capacity (FVC) is the total amount of air that can be exhaled by the patient after a full inhalation. The FVC was measured via spirometry conducted according to internationally accepted standards at 5 min-4 hr post dose of day 1 and week 6.
Time Frame: 5min-4hr at day 1 and week 6 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 + Placebo to Tiotropium | Tiotropium + Placebo to QVA149 | Placebo
Number analyzed (Participants) | 223 | 220 | 218
Liters
  Day 1 (n=210,219,217) | 3.340 (0.0190) | 3.249 (0.0191) | 3.020 (0.0191)
  Week 6 (n= 205,209,206) | 3.393 (0.0254) | 3.269 (0.0253) | 2.957 (0.0253)

5. Secondary Outcome: Change From Baseline in The Capacity of Daily Living During the Morning (CDLM) Score Averaged Over 6 Weeks of Treatment
Description: The Capacity of Daily Living during the Morning (CDLM) is a self-administered daily assessment. The CDLM asks COPD patients to (i) report their ability to carry out 6 morning activities and (ii) rate the difficulty in performing those activities on a five point Likert-type scale ranging from "not at all difficult" to "extremely difficult". For each of the six morning activities a score ranging from 0 (=so difficult that they could not carry out the activity by themselves) to 5 (not at all difficult to carry out the activity by themselves) is calculated by using the responses from the two questions for each activity. Daily CDLM is calculated using the scores average from the 6 morning activities. CDLM is calculated as the average daily CDLM score over 6 weeks of treatment. The change from baseline in CDLM score over 6 weeks is analyzed using a MIXED model with baseline CDLM score as a covariate. A CDLM score of 0.20 is considered to be a minimal clinically important difference.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | QVA149 + Placebo to Tiotropium | Tiotropium + Placebo to QVA149 | Placebo
Number analyzed (Participants) | 167 | 173 | 164
Units on a scale | 0.09 (0.020) | 0.08 (0.020) | -0.01 (0.020)

6. Secondary Outcome: Change From Baseline in the Mean Daily Number of Puffs of Rescue Medication Used Over the 6 Weeks of Treatment
Description: The number of puffs of rescue medication taken by participants, were collected each day during the study via entries in e-diaries
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: puffs
Arm/Group | QVA149 + Placebo to Tiotropium | Tiotropium + Placebo to QVA149 | Placebo
Number analyzed (Participants) | 212 | 215 | 206
puffs | -1.02 (0.202) | -0.57 (0.202) | 0.41 (0.203)

ADVERSE EVENTS:
Arm/Group | QVA149 + Placebo to Tiotropium | Tiotropium + Placebo to QVA149 | Placebo
Serious Adverse Events (participants affected / at risk) | 6/223 | 6/220 | 5/218
Other Adverse Events (participants affected / at risk) | 51/223 | 58/220 | 70/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 + Placebo to Tiotropium (N=223) | Tiotropium + Placebo to QVA149 (N=220) | Placebo (N=218)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Pleural infection bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 + Placebo to Tiotropium (N=223) | Tiotropium + Placebo to QVA149 (N=220) | Placebo (N=218)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Fatigue (General disorders) | 0 | 4 | 3
Influenza like illness (General disorders) | 2 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 4
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 14 | 8 | 13
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 4
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Headache (Nervous system disorders) | 2 | 6 | 3
Sciatica (Nervous system disorders) | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 | 19 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Hypertension (Vascular disorders) | 3 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.